CLINICAL TRIAL: NCT06552572
Title: Phase II Study of Glofitamab Therapy in Relapsed or Refractory Diffuse Large B-cell Lymphoma Patients Achieving Response After CD19 Chimeric Antigen Receptor T-cell Therapy
Brief Title: Glofitamab in Relapsed or Refractory Diffuse Large B-cell Lymphoma After CD19 Chimeric Antigen Receptor T-cell Therapy
Acronym: Glory
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO44989
Record Dates: First submitted 2024-08-03; First posted 2024-08-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; Glofitamab; CD19 CAR T-cell
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab

STUDY DESIGN:
Intervention Model Description: Patients with relapsed or refractory diffuse large B-cell lymphoma who respond to CD19 CAR T-cell therapy: Partial response at one or three months after CAR T-cell therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Glofitamab (Experimental): Glofitamab every 21 days for 12 cycles or until progression.
  1. First cycle
     * Obinutuzumab (GPT) 1000mg (D1)
     * Glofitamab step up dosing 2.5mg (D8) → 10mg (D15)
  2. After the first cycle (completed priming): 30mg IV every 3 weeks.
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab is administered to patients who have residual disease after CD19 CAR T-cell therapy for their relapsed or refractory diffuse large B-cell lymphoma
  Other Names: Columvi® (Roche)

SUMMARY:
The objective of this clinical trial is to determine whether the CD20-CD3 bispecific antibody, glofitamab, is effective in treating residual diffuse large B-cell lymphoma (DLBCL) in adults who have responded to CD19 Chimeric antigen receptor (CAR) T-cell therapy for their relapsed or refractory DLBCL. Additionally, the trial will assess the safety of glofitamab in patients undergoing CD19 CAR T-cell therapy. The primary questions to be addressed are:

Does glofitamab reduce the number of participants experiencing disease progression following CD19 CAR T-cell therapy? What are the medical complications in participants already treated with CD19 CAR T-cell therapy when administered glofitamab?

Participants are required to:

Receive glofitamab every 21 days for 12 cycles or until disease progression. Attend the clinic for checkups and tests every three weeks.

DETAILED DESCRIPTION:
1. Background CD19 CAR T-cell therapy has proven to be a highly effective adoptive cell therapy, evidenced by the significant complete response rates in patients with B-cell acute lymphoblastic leukemia (B-ALL) and large B-cell lymphoma (DLBCL), leading to FDA approvals. While CAR-T cell therapy has been a lifeline for patients unresponsive to other treatments, 60% still experience disease progression despite 40% achieving a complete response. The durability of remission may be compromised by factors such as loss of the target antigen CD19, inhibitory receptor expression, absence of costimulatory ligands, limited CAR-T cell expansion or persistence, and impaired effector function due to exhaustion. Glofitamab, a novel bispecific T-cell engaging antibody, binds bivalently to CD20 on B-cells and monovalently to CD3 on T-cells. Pharmacodynamic studies show that glofitamab administration leads to T-cell activation, indicated by increased granzyme B expression, suggesting it may alter the tumor immune environment towards T-cell activation. We hypothesize that glofitamab could bridge the gap between CAR T- or cytotoxic cells and tumor cells, mitigating immune exhaustion. This could potentially enhance survival by preventing immune cell exhaustion and boosting the efficacy of immunotherapy. Therefore, we aim to conduct a prospective study to augment the therapeutic efficacy of CAR-T cells by bolstering effector cells within the tumor immune environment, using glofitamab as a subsequent treatment post-CAR-T cell therapy.
2. Study population

   * Patients who show partial response at 1 or 3 months after CD19 CAR T-cell therapy for thier relapsed or refractory DLBCL (RR-DLBCL)
3. Treatment protocol A) Glofitamab every 21 days for 12 cycles or until progression.

   1. First cycle

      * Obinutuzumab (GPT) 1000mg (D1)
      * Glofitamab step up dosing 2.5mg (D8) → 10mg (D15)
   2. After the first cycle (completed priming)

      * Glofitamab 30mg IV every 3 weeks B) Supportive care
      * Concomitant administration is recommended during the period of glofitamab administration. Changes in dose and duration are at the decision of the investigators.
      * TMP-SMX 400/800mg QD
      * Acyclovir 200-400mg QD
4. Sample sixe - Previous phase II clinical trials of Tixacel associated a treatment response rate of 40-52% in RR-DLBCL, a 1-year progression-free survival (PFS) of 33%-44%, and a 2-year PFS of 31-36% [5, 6 ]. The new maintenance treatment group used a better effect than the previous physiotherapy treatment and Tixacel treatment alone, setting everyone up. Therefore, the measurement range: H0 S0=S1 vs H1: S0≠S1; S0, S1: According to the definition as the 1-year PFS of the Historical Control group (S0) and the test group (S1), the 1-year PFS of the Historical Control group was 37%, power 90%, law level 5%, training period 2 years, follow-up Assuming that the period of 1 year and the survival time group are exponential, under the hypothesis, the 1-year PFS of the test group is set to 60%, the number of subjects is 28, and the expected event occurrence is 18. With a dropout rate of 5%, the final number of registered participants is 30.

ELIGIBILITY:
A) Inclusion Criteria:

1. Signed informed consent form.
2. Age ≥ 18 years at the time of signing the informed consent form.
3. Histologically diagnosed diffuse large B-cell lymphoma, NOS initially, as defined by 2016 WHO guidelines and confirmed relapsed and refractory disease, defined as follows.

   * Relapsed: the disease that has recurred following a response that lasted over 6 months after completing the last line of therapy.
   * Refractory: the disease that did not respond to or that progressed less than 6 months after completion of the last line of therapy
4. RR-DLBCL patients who should undergo CD 19 CAR-T cell treatment prior to recruitment of this study have achieved partial response (PR) at one or three months after CAR-T cell infusion (If the patient achieves PR at one or three months, patients have to enroll within at least 3 months after CAR-T cell infusion.)
5. ECOG PS: 0-2
6. Adequate hematologic function, as defined by the following laboratory values (If cytopenia is associated with bone marrow involvement, the subject is excluded):

   * Absolute neutrophil > 1,000/mm3
   * Hemoglobin > 9.0 g/dL (Transfusion free within 21 days prior to administration of glofitamab)
   * Platelet > 75,000/mm3 (Transfusion free within 21 days prior to administration of glofitamab)
   * If the patient does not recover neutropenia at one month even though achieving PR, the investigator could wait until 3 months from first achieving PR at one month. However, the patient has to remain in PR status.
7. Negative SARS-CoV-2 antigen or PCR test within 7 days prior to enrollment
8. Adequate organ function, as defined by the following laboratory values

   * AST, ALT < 3.0x upper limit of normal (ULN).
   * Total bilirubin < 1.5 X ULN(Patients with a documented history of Gilbert's Syndrome and in whom total bilirubin elevations are accompanied by elevated indirect bilirubin are eligible if the total bilirubin is ≤ 3x ULN).
   * Serum creatinine ≤ 1.5 mg/dL, Creatinine clearance ≥ 50ml/min.
9. Female subjects are required to meet the following criteria:

   * Pregnancy test: For women of childbearing potential, a negative serum or urine pregnancy test at screening
   * Contraception: Patients must agree to either remain completely abstinent or to use two effective contraceptive methods that result in a failure rate of < 1% per year from screening; until at least 3 months after pre-treatment with obinutuzumab, 2 months after the last dose of glofitamab, 2 months after the last dose of tocilizumab (if applicable), whichever is longer if the patient is a male. If the patient is female, effective contraception should be used until at least 18 months after pre-treatment with obinutuzumab, 2 months after the last dose of glofitamab, or 3 months after the last dose of tocilizumab (if applicable), whichever is longer.( Men must refrain from donating sperm during this same period)
10. Male subjects are required to meet the following criteria

    * With a female partner of childbearing potential or pregnant female partners, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year for at least 6 months after the last dose of the study treatment.
    * Men must refrain from donating sperm during this study period.
11. Having tumor tissue samples in storage available for targeted sequencing
12. At least one bi-dimensionally measurable (≥ 1.5 cm) nodal lesion, or one bi-dimensionally measurable (≥1 cm) extranodal lesion, as measured on CT scan
13. Life expectancy ≥ 12 weeks

B) Exclusion Criteria:

1. Patients have failed to respond to CD19 CAR-T cell therapy.
2. Patients who received previously treated bispecific antibodies.
3. Current or past history of primary or secondary central nervous system (CNS) lymphoma.
4. Peripheral neuropathy was assessed to be grade >1 according to NCI CTCAE v5.0 at enrollment.
5. Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease.

   - Patients with a history of stroke who have not experienced a stroke of transient ischemic attack within the past 2 years and have no residual neurologic deficits, as judged by the investigator, are allowed.
6. Any of the following abnormal laboratory values, unless abnormal laboratory values are associated with the underlying lymphoma per the investigator. (Patients with a documented history of Gilbert's Syndrome and in whom total bilirubin elevations are accompanied by elevated indirect bilirubin are eligible if the total bilirubin is ≤ 3 × ULN)

   * AST/ ALT ≥ 3.0 X upper limit of normal (ULN).
   * Total bilirubin ≥ 1.5 X ULN.
7. Has a concomitant malignancy or had a malignancy (except for appropriately treated basal or squamous cell carcinoma or cervical carcinoma in situ) in the last 3 years prior to initiation of the study treatment
8. Underwent a major surgery within 21 days prior to initiating the study treatment or has not recovered from severe side effects of surgery
9. Concomitant use of immunosuppressants, except for the following:

   - Intranasal, inhaled, or topical steroid, or local steroid injection (such as intra-articular injection)
   * Physiological dose ≤ 10 mg/day of prednisone or equivalent doses of systemic corticosteroid
   * Premedication with steroids to prevent hypersensitivity reaction (such as premedication prior to a CT scan). At the discretion of the investigator, the use of prednisolone at ≥10 mg for adrenal insufficiency may be acceptable.
10. Clinically significant or active cardiovascular disease

    * Myocardial infarction: within 6 months prior to study entry
    * Unstable angina, congestive heart failure (New York Heart Association class ≥III) or Objective Assessment Class C or D cardiac disease, or serious cardiac arrhythmias requiring medication, including any of the following: ➀ Left ventricular ejection fraction (LVEF) < 50% as measured by echocardiography, ➁ QTc > 480 msec (using the QTcF formula) on ECG at screening, ➂ unstable angina, ④ ventricular arrhythmias except for benign premature ventricular contractions, ⑤ medically uncontrolled supraventricular and nodal arrhythmias, ⑥ conduction abnormality requiring a pacemaker, ⑦ valve disease with documented cardiac dysfunction
11. Other concomitant severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes mellitus, chronic pancreatitis, active chronic hepatitis, etc.) that the investigator considers would preclude the subject's participation in the clinical trial.

    * Other severe acute or chronic medical conditions include colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis, or psychiatric conditions, including recent (in the last 1 year) or active suicidal thoughts or behaviors; or laboratory abnormalities that, in the investigator's opinion, may increase the risk associated with participation in the clinical trial or study treatment, or that may interfere with the interpretation of clinical trial results.
12. Active infection or reactivation of a latent infection, whether bacterial, viral (including, but not limited to SARS-COV-2, EBV, cytomegalovirus (CMV), hepatitis B, hepatitis C, and HIV), fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or requiring systemic therapy within 4 weeks prior to the first study drug infusion.
13. Active autoimmune diseases may be exacerbated upon administration of immunostimulants.

    - However, subjects with type I diabetes mellitus, vitiligo, psoriasis, or hypothyroidism, or hyperthyroidism not requiring immunosuppressive treatment are eligible.
14. Incapable of understanding or complying with clinical trial instructions and requirements or have a history of noncompliance with medical therapy
15. Pregnant or nursing (breastfeeding) women.

    - Pregnancy is defined as the condition of a woman from pregnancy as confirmed by positive serum hCG laboratory test (>5 mIU/mL) to termination of pregnancy.
16. Live vaccination is prohibited within 4 weeks prior to the first dose and during clinical trial participation.

    * However, inactivated vaccines such as, influenza and COVID vaccines are allowed.
    * Concomitant administration of an approved non-live COVID-19 vaccine is permitted. Examples of permitted vaccines include mRNA, inactivated virus, and replication-deficient viral vector vaccines. The decision on whether and when to administer a COVID-19 vaccine should be individualized by the investigator in consultation with the patient.
    * Factors to consider when making the individualized decision for patients receiving glofitamab include the following:

      * Risk of SARS-CoV-2 infection and potential benefit from the vaccine
      * The general condition of the patient and potential complications associated with SARS-CoV-2 infection
      * Severity and seriousness of the underlying disease
      * Epidemiology of COVID-19 in the Patient's Location
    * For patients who plan to receive a COVID-19 vaccine that requires two doses, it is recommended they complete the course of vaccination (i.e., they should receive the second dose) at least seven days before starting study treatment in order to maximize vaccine efficacy. For vaccines that require a single dose, patients are recommended to be vaccinated at least 28 days before starting study therapy in order to maximize vaccine efficacy unless a delay in treatment is clinically unacceptable.
    * If a COVID-19 vaccine is administered while the patient is already receiving treatment with glofitamab, the COVID-19 vaccine should be administered in the middle of a treatment cycle, for example, one week before or after a dose of glofitamab. The administration of the vaccine should be timed to take place after the completion of the glofitamab step-up dosing and at least one week after the administration of the target glofitamab dose.
    * Cytokine-release syndrome (CRS) is a risk for glofitamab that occurs most commonly during step-up dosing. Many COVID-19 vaccines are highly immunogenic, and their risk of potentiating CRS is unknown.
17. Hepatitis B virus (HBV) related liver disease, such as the following:

    * Chronic hepatitis with cirrhosis
    * HBV reactivation (Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable, provided that they are willing to undergo DNA testing on Day 1 of every cycle and every 3 months for at least 12 months after the last cycle of study treatment and appropriate antiviral therapy.)
    * Hepatitis B virus (HBV) infection at screening (HBV surface antigen-positive and HBV DNA-positive)
18. Hepatitis C virus (HCV) infection at screening (HCV RNA positive if positive for anti-HCV antibody at screening)

    - Positive test results for hepatitis C virus (HCV) antibody - Patients who are positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
19. Known history of human immunodeficiency virus (HIV) seropositive status; for patients with unknown HIV status, HIV testing will be performed at screening.

    - Individuals with a positive HIV test at screening are eligible, provided they are stable on antiretroviral therapy, have a CD4 count ≥ 200/μL, and have an undetectable viral load. HIV positive patients should be monitored per local/institutional standards while receiving study treatment.
20. Positive SARS-CoV-2 infection within 30 days prior to the first study treatment, including asymptomatic SARS-CoV-2 infection.

    - Patients may be eligible if they have no persistent respiratory symptoms, no evidence of lung infiltrates on chest CT, and have a negative PCR during the 30 days prior to the first study treatment.
21. Known or suspected chronic active Epstein-Barr virus infection.
22. Prior solid organ transplantation.
23. Prior allogeneic stem cell transplantation.
24. History of Progressive multifocal leukoencephalopathy (PML).
25. Known or suspected history of HLH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year progression free survival rate after enrollment | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years
  Measurement of progression-free survival after CD19 CAR T-cell therapy

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years
  Hematological and non-hematological toxicities associated with glofitamab therapy

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD., PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No